CLINICAL TRIAL: NCT00322049
Title: A Phase I/II Trial of Tetravalent Live Attenuated Dengue Vaccine in Flavivirus Antibody Naive Infants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WRAIR 824; HSRRB Log A-10064 (Other: USAMRMC); GSK CPMS7663310/001 (Other: GSK); DEN-001 (Other: GSK)
Record Dates: First submitted 2006-05-03; First posted 2006-05-04 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: Dengue
Keywords: Dengue, Vaccine, Thailand
MeSH Terms: conditions — Dengue | interventions — Chickenpox Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A: Dengue Vaccine- Full Dose (T-DEN F17 ) (Experimental): Dengue vaccine at Months 0 and 6 and booster follow-up at 3 years;
  DEN candidate vaccine: One dose of the tetravalent, live attenuated DEN vaccine candidate, F17, contains dengue serotype 1, 2, 3 and 4 vaccines. This formulation contains 50 mcg/mL neomycin base, 5.5% lactose, and 1.9 g/dL human serum albumin; for subcutaneous injection. All infants subsequently received an inactivated JE vaccine approximately one and 1.5 months following dengue vaccine dose 2. The licensed JE vaccine in liquid form, was dosed at 0.25 ml for subcutaneous injection.
  Interventions: Biological: Tetravalent live attenuated dengue vaccine
- Cohort B: Control vaccines (Active Comparator): Control vaccines: Hemophilus influenza type b (Hib) vaccine and varicella vaccine
  Interventions: Biological: Varicella vaccine and Haemophilus influenzae Type b Conjugate vaccine
- Cohort C: Dengue Vaccine - 1/10 Dose (T-DEN F17 ) (Experimental): Dengue vaccine at Months 0 and 6 and booster follow-up at 3 years
  Interventions: Biological: Tetravalent live attenuated dengue vaccine

INTERVENTIONS:
Biological: Tetravalent live attenuated dengue vaccine — DEN candidate vaccine: One dose of the tetravalent, live attenuated DEN vaccine candidate, F17, contains dengue serotype 1, 2, 3 and 4 vaccines. This formulation contains 50 mcg/mL neomycin base, 5.5% lactose, and 1.9 g/dL human serum albumin; for subcutaneous injection.
  Infants received dengue vaccine at study months 0 and 6 or control vaccine (varicella vaccine at study month 0 and Haemophilus influenzae Type b Conjugate vaccine at study month 6). Both control vaccines are licensed for use in Thailand.
  All infants subsequently received an inactivated JE vaccine approximately one and 1.5 months following dengue vaccine dose 2. The licensed JE vaccine in liquid form, was dosed at 0.25 ml for subcutaneous injection.
  A booster dose of DEN vaccine was given to all subjects previously vaccinated with DEN vaccine in Dengue -001. The booster dose was administered approximately 42 months after dose 2 (at the Year 3 visit).
  Arms: Cohort A: Dengue Vaccine- Full Dose (T-DEN F17 ); Cohort C: Dengue Vaccine - 1/10 Dose (T-DEN F17 )
Biological: Varicella vaccine and Haemophilus influenzae Type b Conjugate vaccine — Infants received dengue vaccine at study months 0 and 6 or control vaccine (varicella vaccine at study month 0 and Haemophilus influenzae Type b Conjugate vaccine at study month 6). Both control vaccines are licensed for use in Thailand.
  Arms: Cohort B: Control vaccines

SUMMARY:
The main target populations for the tetravalent live attenuated dengue virus vaccine are indigenous populations, especially infants less than 2 years old, residing in areas of the world endemic for dengue and at risk of developing dengue hemorrhagic fever (DHF). The presence of maternal dengue antibody during the first year of life makes it unlikely that a vaccine given during that time will have long-term efficacy, as the vaccine virus would likely be neutralized prior to necessary replication. Children older than 18 months may have preexisting flavivirus antibody. Therefore, vaccination of infants living in Thailand early in the second year of life (between the ages of 12 and 18 months) seems most beneficial. The aim of this trial is to evaluate the safety and immunogenicity of a two-dose schedule of a tetravalent live attenuated dengue vaccine in flavivirus antibody naïve infants beginning at 12-15 months of age.

* To assess the kinetics of dengue neutralizing antibodies to each dengue virus serotype one and four years following dose 2 of dengue/control vaccination in the setting of potential wild-type dengue virus exposure.
* To assess the immunogenicity, the safety and reactogenicity of a booster dose of dengue vaccine administered at Year 3 following primary vaccination.

DETAILED DESCRIPTION:
* This is a Phase I/II, randomized, observer-blind, controlled trial. Thirty-four flavivirus naïve infants will be randomized to the vaccine group and 17 infants to the control group.
* Infants receive dengue vaccine at study months 0 and 6 or control vaccine (Varicella vaccine at study month 0 and Haemophilus influenzae Type b Conjugate vaccine at study month 6). Both are licensed for use in Thailand.
* All infants subsequently receive an inactivated JE vaccine approximately one and 1.5 months following dengue vaccine dose 2.
* Infants are monitored daily for 21 days following each dengue or control vaccination and 7 days after each JE vaccination for solicited adverse events. Unsolicited events will be recorded up to 31 days (days 0-30) after dengue/control vaccinations and each day after dose 1 of JE vaccine until the concluding study visit.
* Study duration (excluding screening) is approximately 8.5 months for each subject.
* Each enrollee is followed a four year period following dose 2 of dengue/control vaccination to assess for dengue-related hospitalizations and dengue antibody kinetics.
* Investigators will administer a 3rd dose of tetravalent dengue vaccine to all subjects who received 2 doses of dengue vaccine (0 and 6 months) during the primary phase of the study. The 3rd dose will be administered 3 years following the primary vaccination series. Peripheral blood mononuclear cells (PBMCs) and sera will be collected at the time of dose 3, and twice again at one month and one year following dose 3 from dengue group subjects.

Investigators will address the following questions:

1. Is a 3rd dose of live virus tetravalent dengue vaccine safe in Thai toddlers/children?
2. Is a 3rd dose of live virus tetravalent dengue vaccine required in toddlers/children to induce optimal immune (neutralizing antibody, cellular mediated immunity) responses?
3. Is there evidence of T and B cell memory following a primary dengue vaccination series (dose 1 and 2)?
4. How does a 3rd dose of live virus tetravalent dengue vaccine impact B and T cell memory?

ELIGIBILITY:
Inclusion Criteria:

* Male and female infants between 12 and 15 months (12 and <16 months) of age at the time of the first dengue vaccination
* Free of obvious health problems as established by medical history and clinical examination before entering into the study. As a marker of nutritional status, an infant's weight to height ratio will be above the 5th percentile compared to the standards for same sex and age children cared for at Phramongkutklao Hospital, Bangkok, Thailand
* Written informed consent obtained from the parent of the subject.

Amendment 8 Inclusion Criteria:

* Completed the Dengue-001 study having previously received 2 doses of experimental dengue vaccine according to protocol.
* Written informed consent obtained from the parent or guardian of the subject. (obtained in amendment 5)
* Written informed consent obtained from the parent or guardian of the subject who agrees to their child's participation to receive a dengue booster dose and booster follow-up.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the protocol-specified vaccines within 30 days preceding the administration of the first dose of dengue/control vaccine or planned use during the study period
* Administration of a registered vaccine within 30 days preceding the first study vaccination or planned administration within 30 days prior to, or 30 days after any protocol-specified vaccine administration
* MMR vaccination given within 60 days prior to the first dose of dengue/control vaccine (added bullet point, or planned administration within 60 days prior to, or 30 days after any protocol-specified vaccine administration
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs during the study period. (For corticosteroids, this will mean prednisone, or equivalent, 0.5 mg/kg/day. Inhaled and topical steroids are allowed.
* Any confirmed or suspected immunosuppressive or immunodeficient condition
* Any clinically significant history, including any seizures or other serious medical condition as determined by the investigator
* A first order family member (parent or sibling) with a history of chronic headaches
* A first order family member (parent or sibling) with a history of a congenital or hereditary immunodeficiency
* Abnormal clinical laboratory screening test results (based on normal values set by the laboratory) that are deemed clinically significant by study investigators and/or the Medical Monitor
* The presence of HBsAg or antibodies against HIV or HCV at screening
* Pre-existing antibody to dengue 1-4 virus serotypes or Japanese encephalitis virus (JEV) by HAI or PRNT50 at screening
* Previous vaccination against yellow fever virus, JEV, tick-borne encephalitis virus (TBE), varicella virus or booster dose of Hib in the second year of life
* History of varicella disease or invasive Haemophilus Influenzae B disease
* Acute disease at time of enrollment (Acute illness is defined as the presence of a moderate or severe illness with or without fever). All vaccines can be administered to persons with a minor illness such as diarrhea or mild upper respiratory infection with or without low-grade febrile illness, i.e., axillary temperature <37.5°C (<99.5°F).
* Administration of immunoglobulins and/or blood products since birth or planned administration during the study period
* Known allergic or idiosyncratic reaction to neomycin or related antibiotics (including streptomycin, gentamicin, amikacin, , tobramycin, kanamycin and bacitracin)
* Allergy to dogs or monkeys or hypersensitivity to proteins of rodent or neural origin
* Allergy to gelatin or hypersensitivity to thimerosal
* Infant whose parent has no easy access to a fixed or mobile telephone
* Parental illiteracy
* Plans to leave Bangkok during the first 8.5 months after initial vaccination or definite plans to move from Bangkok during the 5 years following first dose dengue/control vaccination.

Amendment 8 Exclusion Criteria:

-Any subject with confirmed dengue hemorrhagic fever during the 2 to 3 year period before booster dose administration will not be eligible for enrollment for the booster.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2004-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert V. Gibbons, MD, Principal Investigator — U.S. Army Medical Component Armed Forces Research Institute of Medical Sciences (USAMC-AFRIMS); Veerachai Watanaveeradej, MD, Principal Investigator — Infectious Disease Department of Pediatrics Phramongkutklao Hospital
Locations (1):
- USAMC-AFRIMS/Department of Pediatrics, Pharamongkutklao Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Watanaveeradej V, Simasathien S, Nisalak A, Endy TP, Jarman RG, Innis BL, Thomas SJ, Gibbons RV, Hengprasert S, Samakoses R, Kerdpanich A, Vaughn DW, Putnak JR, Eckels KH, Barrera Rde L, Mammen MP Jr. Safety and immunogenicity of a tetravalent live-attenuated dengue vaccine in flavivirus-naive infants. Am J Trop Med Hyg. 2011 Aug;85(2):341-51. doi: 10.4269/ajtmh.2011.10-0501. PMID 21813857

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 51 infants enrolled and vaccinated for safety cohort, all received dose 1 and 50 completed the study. 49 vaccinated for ATP immunogenicity cohort.
Groups:
- Cohort A - 1/10th Dose Dengue Vaccine: 1/10th full dose at study months 0 and 6 or control vaccines (varicells vaccine at study month 0 and Hib vaccine at study month 6)
- Cohort B - Full Dose Dengue Vaccine: Full-dose of dengue vaccine at study months 0 and 6 or control vaccines (varicells vaccine at study month 0 and Hib vaccine at study month 6)
- Cohort C - Full Dose Dengue Vaccine: Full-dose dengue vaccine at study months 0 and 6 or control vaccines (varicells vaccine at study month 0 and Hib vaccine at study month 6)
- Control Group - Hib Vaccine: Hemophilus influenza type b (Hib) vaccine and varicella vaccine
Period: Overall Study
Arm/Group | Cohort A - 1/10th Dose Dengue Vaccine | Cohort B - Full Dose Dengue Vaccine | Cohort C - Full Dose Dengue Vaccine | Control Group - Hib Vaccine
Started | 4 | 10 | 20 | 17
Completed | 4 | 9 | 20 | 16
Not Completed | 0 | 1 | 0 | 1
Not completed — Moved out of area | 0 | 0 | 0 | 1
Not completed — Infected with Dengue during study | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - 1/10th Dose Dengue Vaccine | Cohort B - Full Dose Dengue Vaccine | Cohort C - Full Dose Dengue Vaccine | Control Group - Hib Vaccine | Total
Number analyzed (Participants) | 4 | 10 | 20 | 17 | 51
Age, Continuous [Mean (Standard Deviation); unit: months] | 14.0 (0.00) | 13.3 (0.82) | 13.6 (0.88) | 13.6 (0.79) | 13.6 (0.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7 | 9 | 23
  Male | 3 | 4 | 13 | 8 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Southeast Asian | 4 | 10 | 20 | 17 | 51
Region of Enrollment [Number; unit: participants]
  Thailand | 4 | 10 | 20 | 17 | 51

OUTCOME MEASURES:

1. Primary Outcome: Reactogenicity in Terms of Solicited Symptoms After Dose 1 of the Dengue Vaccine vs. Control Vaccine.
Description: Local and general solicited reactogenicity using diary cards for 21 days (days 0-20) after the first dose of dengue/control vaccine
Time Frame: 21-day follow-up period after Dose 1
Population: Format of results is consistent with how data was presented in the Final Clinical Study Report. Combining of cohorts B and C was due to both cohorts being full dose
Measure: Number; unit: specified events
Groups:
- Cohorts B & C - Full Dose Dengue Vaccine: Full-dose of dengue vaccine at study months 0 and 6 or control vaccines (varicells vaccine at study month 0 and Hib vaccine at study month 6)
Arm/Group | Control Group - Hib Vaccine | Cohort A - 1/10th Dose Dengue Vaccine | Cohorts B & C - Full Dose Dengue Vaccine
Number analyzed (Participants) | 17 | 4 | 30
specified events
  Dose 1 : Pain | 3 | 1 | 11
  Dose 1 : Redness | 1 | 2 | 21
  Dose 1 : Swelling | 2 | 1 | 16
  Dose 2 : Pain | 2 | 1 | 13
  Dose 2 : Redness | 3 | 1 | 13
  Dose 2 : Swelling | 1 | 1 | 8
  Overall / dose : Pain | 5 | 2 | 24
  Overall / dose : Redness | 4 | 3 | 34
  Overall / dose : Swelling | 3 | 2 | 24
  Overall / subject : Pain | 3 | 1 | 18
  Overall / subject : Redness | 3 | 2 | 22
  Overall / subject : Swelling | 2 | 1 | 19
  Overall / dose - Cough | 15 | 4 | 27
  Overall / dose - Decreased activity | 11 | 2 | 11
  Overall / dose - Drowsiness | 12 | 0 | 18
  Overall / dose - Irritability | 13 | 3 | 23
  Overall / dose - Loss of appetite | 13 | 2 | 21
  Overall / dose - Fever (axillary celsius) | 16 | 3 | 24
  Overall / dose - Vomiting | 12 | 2 | 24

2. Primary Outcome: Geometric Mean Titers (GMT) for N Antibody to All Four Serotypes and Japanese Encephalitis (JE) Vaccine
Description: Assess the immunogenicity of the dengue vaccine in terms of GMTs 30 days post-Dose 2 of dengue vaccine for all four serotypes (DEN-1, 2, 3, 4 and JE (Japanese encephalitis)). Analysis of immunogenicity was performed on the ATP cohort.
Time Frame: 30 days post Dose 2
Population: GMT calculated on all subjects. Dil = Dilution; P1(M1) = blood sampling on month after dose 1, at study month 1; PII(M7) = blood sampling one month after dose 2, at study month 7; PII(M8.5) = blood sampling 2 1/2 months after dose 2, at study month 8.5. Combining of cohorts B and C was due to both cohorts being full dose
Measure: Mean (95% Confidence Interval); unit: titers
Arm/Group | Control Group - Hib Vaccine | Cohort A - 1/10th Dose Dengue Vaccine | Cohorts B & C - Full Dose Dengue Vaccine
Number analyzed (Participants) | 17 | 4 | 30
titers
  DEN-1 GMT - PI(M1) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.2 [4.8 to 5.5]
  DEN-1 GMT - PII(M7) | 5.0 [5.0 to 5.0] | 6.1 [3.3 to 11.4] | 20.7 [11.4 to 37.7]
  DEN-2 GMT - PI(M1) | 5.0 [5.0 to 5.0] | 8.8 [1.4 to 54.4] | 13.7 [7.7 to 24.5]
  DEN-2 GMT - PII(M7) | 5.0 [5.0 to 5.0] | 173.6 [50.1 to 601.5] | 239.6 [163.6 to 351.1]
  DEN-3 GMT - PI(M1) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  DEN-3 GMT PII(M7) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 29.2 [18.6 to 45.7]
  DEN-4 GMT PI(M1) | 5.0 [5.0 to 5.0] | 15.7 [0.4 to 600.1] | 22.5 [10.0 to 50.3]
  DEN-4 GMT PII(M7) | 5.0 [5.0 to 5.0] | 31.9 [2.5 to 408.2] | 52.5 [29.0 to 95.0]
  JE Vaccine GMT PI(M1) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 6.0 [5.0 to 7.2]
  JE Vaccine GMT PII(M7) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 8.3 [5.1 to 13.6]
  JE Vaccine GMT PII(M8.5) | 16.8 [7.4 to 38.1] | 19.3 [7.0 to 52.9] | 12.9 [6.7 to 24.6]

3. Primary Outcome: Percent of Participants With Seronegative Neutralizing (N) Antibody Titers to Each DEN Serotype After Dose 2
Description: Seronegative for N antibody against DEN 1, 2, 3 and 4 antibody after dengue dose 2.
  Seronegative (antibody titer <10 1/Dil for N lg to DEN-1, N lg to DEN-2, N lg to DEN-3, N lg) prior to vaccination.
Time Frame: month 7 after dose 2
Measure: Mean (95% Confidence Interval); unit: % of responders
Groups:
- Cohorts B & C - Full Dose Dengue Vaccine: Full dose dengue vaccine at study months 0 and 6
Arm/Group | Cohort A - 1/10th Dose Dengue Vaccine | Cohort B - Full Dose Dengue Vaccine | Cohort C - Full Dose Dengue Vaccine | Cohorts B & C - Full Dose Dengue Vaccine
Number analyzed (Participants) | 4 | 9 | 20 | 29
% of responders
  N lg to DEN-1 (Dil) | 25.0 [0.6 to 80.6] | 88.9 [51.8 to 99.7] | 40.0 [19.1 to 63.9] | 55.2 [35.7 to 73.6]
  N lg to DEN-2 (Dil) | 100 [39.8 to 100] | 100 [66.4 to 100] | 100 [82.4 to 100] | 100 [87.7 to 100]
  N lg to DEN-3 (Dil) | 0.0 [0.0 to 0.0] | 100 [66.4 to 100] | 80.0 [56.3 to 94.3] | 86.2 [68.3 to 96.1]
  N lg to DEN-4 (Dil) | 75.0 [19.4 to 99.4] | 100 [66.4 to 100] | 94.7 [74.0 to 99.9] | 96.4 [81.7 to 99.9]

4. Primary Outcome: Percent of Participants With Seronegative Neutralizing (N) Antibody Titers to Each DEN Serotype After Dengue Dose 2 (and 2 Doses of JE
Description: Seropositivity for N antibody against DEN 1, 2, 3 and 4 antibody after dengue dose 2 (and 2 doses of JE).
  Seronegative (antibody titer <10 1/Dil for N lg to DEN-1, N lg to DEN-2, N lg to DEN-3, N lg) prior to vaccination.
Time Frame: month 8.5
Measure: Mean (95% Confidence Interval); unit: % of responders
Arm/Group | Cohort A - 1/10th Dose Dengue Vaccine | Cohort B - Full Dose Dengue Vaccine | Cohort C - Full Dose Dengue Vaccine | Cohorts B & C - Full Dose Dengue Vaccine
Number analyzed (Participants) | 4 | 9 | 20 | 29
% of responders
  N lg to DEN-1 (Dil) | 25.0 [0.6 to 80.6] | 55.6 [21.2 to 86.3] | 35.0 [15.4 to 59.2] | 41.4 [23.5 to 61.1]
  N lg to DEN-2 (Dil) | 100 [39.8 to 100] | 100 [66.4 to 100] | 100 [82.4 to 100] | 100 [87.7 to 100]
  N lg to DEN-3 (Dil) | 25.0 [0.6 to 80.6] | 77.8 [40.0 to 97.2] | 60.0 [36.1 to 80.9] | 65.5 [45.7 to 82.1]
  N lg to DEN-4 (Dil) | 50.0 [6.8 to 93.2] | 88.9 [51.8 to 99.7] | 60.0 [36.1 to 80.9] | 69.0 [49.2 to 84.7]

5. Primary Outcome: JE Vaccine Response
Description: Seropositivity rates and GMTs for N lg to JEV antibodies. Pre= Pre vaccination, blood sampling prior to the first vaccine dose; PI(M1)= Post 1, month 1, blood sampling one month after dose 1 at study month 1; PI(M6)= Post 1, month 6, blood sampling 6 months after dose 1 at study month 6; PII(M7)= Post II, month 7, blood sampling one month after dose 2 at study month 7; PIV(M8.5)= Post IV, month 8.5, blood sampling after 2 doses of dengue/control and 2 doses of JE vaccines at study month 8.5
Time Frame: Pre-vaccination, 1, 6, 7 and 8.5 months after two doses of dengue vaccine
Population: Combining of cohorts B and C was due to both cohorts being full dose
Measure: Mean (95% Confidence Interval); unit: % of subjects with titer within range
Arm/Group | Control Group - Hib Vaccine | Cohort A - 1/10th Dose Dengue Vaccine | Cohorts B & C - Full Dose Dengue Vaccine
Number analyzed (Participants) | 16 | 4 | 29
% of subjects with titer within range
  N lg against JEV >10 1/Dil - PRE | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 11.9]
  GMT - PRE | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  N lg against JEV >10 1/Dil - PI(M1) | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 60.2] | 13.8 [3.9 to 31.7]
  GMT - PI(M1) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 6.0 [5.0 to 7.2]
  N lg against JEV >10 1/Dil - PI(M6) | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 11.9]
  GMT - PI(M6) | 5.3 [4.7 to 5.9] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  N lg against JEV >10 1/Dil - PII(M7) | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 60.2] | 17.9 [6.1 to 36.9]
  GMT - PII(M7) | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 8.3 [5.1 to 13.6]
  N lg against JEV >10 1/Dil - PIV(M8.5) | 56.3 [29.9 to 80.2] | 100 [39.8 to 100] | 32.1 [15.9 to 52.4]
  GMT - PIV(M8.5) | 16.8 [7.4 to 38.1] | 19.3 [7.0 to 52.9] | 12.9 [6.7 to 24.6]

6. Secondary Outcome: Incidence of Dengue Specific Symptoms
Description: Percentage of subjects showing incidence of dengue specific symptoms during the 30-day follow-up period after vaccinations
Time Frame: 30-day follow-up period after dose 1 and 2
Measure: Mean (95% Confidence Interval); unit: % of subjects with specified symptoms
Groups:
- Control Group: Hemophilus influenza type b (Hib) vaccine and varicella vaccine
Arm/Group | Control Group | Cohort A - 1/10th Dose Dengue Vaccine | Cohort B - Full Dose Dengue Vaccine | Cohort C - Full Dose Dengue Vaccine | Cohorts B & C - Full Dose Dengue Vaccine
Number analyzed (Participants) | 17 | 4 | 10 | 20 | 30
% of subjects with specified symptoms
  Dose 1 - Rash | 5.9 [0.15 to 28.69] | 0.0 [0.00 to 60.24] | 30.0 [6.67 to 65.25] | 15.0 [3.21 to 37.89] | 20.0 [7.71 to 38.57]
  Dose 1 - Hemorrhage | 0.0 [0.00 to 19.51] | 0.0 [0.00 to 60.24] | 0.0 [0.00 to 30.85] | 0.0 [0.00 to 16.84] | 0.0 [0.00 to 11.57]
  Dose 1 - Conjunctival hemorrhage | 0.0 [0.00 to 19.51] | 0.0 [0.00 to 60.24] | 0.0 [0.00 to 30.85] | 0.0 [0.00 to 16.84] | 0.0 [0.00 to 11.57]
  Dose 1 - Conjunctival injection | 0.0 [0.00 to 19.51] | 0.00 [0.00 to 60.24] | 0.0 [0.00 to 30.85] | 0.0 [0.00 to 16.84] | 0.0 [0.00 to 11.57]
  Dose 1 - Mucosal hemorrhage | 0.0 [0.00 to 19.51] | 25.0 [0.63 to 80.59] | 0.0 [0.00 to 30.85] | 0.0 [0.00 to 16.84] | 0.0 [0.00 to 11.57]
  Dose 1 - Lymphadenopathy | 70.6 [44.04 to 89.69] | 50.0 [6.76 to 93.24] | 80.0 [44.39 to 97.48] | 50.0 [27.20 to 72.80] | 60.0 [40.60 to 77.34]
  Dose 1 - Hepatomegaly | 0.0 [0.00 to 19.51] | 0.0 [0.00 to 60.24] | 0.0 [0.00 to 30.85] | 0.0 [0.00 to 16.84] | 0.0 [0.00 to 11.57]
  Dose 1 - Splenomegaly | 0.0 [0.00 to 19.51] | 0.0 [0.00 to 60.24] | 0.0 [0.00 to 30.85] | 0.0 [0.00 to 16.84] | 0.0 [0.00 to 11.57]
  Dose 2 - Rash | 11.8 [1.46 to 36.44] | 0.0 [0.00 to 60.24] | 10.0 [0.25 to 44.50] | 5.0 [0.13 to 24.87] | 6.7 [0.82 to 22.07]
  Dose 2 - Hemorrhage | 0.0 [0.00 to 19.51] | 0.0 [0.00 to 60.24] | 0.0 [0.00 to 30.85] | 0.0 [0.00 to 16.84] | 0.0 [0.00 to 11.57]
  Dose 2 - Conjunctival hemorrhage | 0.0 [0.00 to 19.51] | 0.0 [0.00 to 60.24] | 0.0 [0.00 to 30.85] | 0.0 [0.00 to 16.54] | 0.0 [0.00 to 11.57]
  Dose 2 - Conjunctival injecgtion | 5.9 [0.15 to 28.69] | 0.0 [0.00 to 60.24] | 0.0 [0.00 to 30.85] | 15.0 [3.21 to 37.89] | 10.0 [2.11 to 26.53]
  Dose 2 - Mucosal hemorrhage | 0.0 [0.00 to 19.51] | 0.0 [0.00 to 60.24] | 0.0 [0.00 to 30.85] | 0.0 [0.00 to 16.84] | 0.0 [0.00 to 11.57]
  Dose 2 - Lymphadenopathy | 58.8 [32.92 to 81.56] | 75.0 [19.41 to 99.37] | 60.0 [26.24 to 87.84] | 25.0 [8.66 to 49.10] | 36.7 [19.93 to 56.14]
  Dose 2 - Hepatomegaly | 0.0 [0.00 to 19.51] | 0.0 [0.00 to 60.24] | 0.0 [0.00 to 30.85] | 0.0 [0.00 to 16.84] | 0.0 [0.00 to 11.57]
  Dose 2 - Spenomegaly | 0.0 [0.00 to 19.51] | 0.0 [0.00 to 60.24] | 0.0 [0.00 to 30.85] | 0.0 [0.00 to 16.84] | 0.0 [0.00 to 11.57]

7. Secondary Outcome: Percentage of Subjects With a Dengue Viremia 10 Days Post Booster Dose
Description: Percentage of subjects with a dengue viremia 10 days after each dose of vaccine.
  RT PCR = Reverse-transcriptase polymerase chain reaction Nested PCR - Nested polymerase chain reaction
  Per protocol, all participants receiving a Dengue Vaccine were combined for Dengue Viremia assessment via RT-PCR and Nested PCR
Time Frame: 10 days after post dose 1 and 2
Population: All participants with evaluable results are reported via RT-PCR and Nested PCR analysis. Scheduled phlebotomy and unscheduled phlebotomy when a subject was ill during the study revealed dengue viremia by RT-/nested PCR, for seven subjects (2 in cohort B and 5 in cohort C).
Measure: Number; unit: % of subjects
Groups:
- Subject With Viremia Measured by: RT-PCR; Subject With Viremia Measured by: Nested PCR: Scheduled phlebotomy and unscheduled phlebotomy when a subject was ill during the study revealed dengue viremia
Arm/Group | Subject With Viremia Measured by: RT-PCR | Subject With Viremia Measured by: Nested PCR
Number analyzed (Participants) | 34 | 34
% of subjects
  10 days post dose 1 | 2.9 | 14.7
  10 days post dose 2 | 0.0 | 5.9

ADVERSE EVENTS:
Time Frame: 8.5 months
Groups:
- Cohort A: Dengue Vaccine- 1/10 Dose (T-DEN F17 ): Dengue vaccine at Months 0 and 6 and booster follow-up at 3 years;
- Cohort B: Full Dose (T-DEN F17 ): Control vaccines: Hemophilus influenza type b (Hib) vaccine and varicella vaccine
- Cohort C: Dengue Vaccine - Full Dose (T-DEN F17 ): Dengue vaccine at Months 0 and 6 and booster follow-up at 3 years
Arm/Group | Cohort A: Dengue Vaccine- 1/10 Dose (T-DEN F17 ) | Cohort B: Full Dose (T-DEN F17 ) | Cohort C: Dengue Vaccine - Full Dose (T-DEN F17 ) | Control Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/10 | 0/20 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/10 | 0/20 | 3/17
Other Adverse Events (participants affected / at risk) | 4/4 | 10/10 | 20/20 | 6/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Dengue Vaccine- 1/10 Dose (T-DEN F17 ) (N=4) | Cohort B: Full Dose (T-DEN F17 ) (N=10) | Cohort C: Dengue Vaccine - Full Dose (T-DEN F17 ) (N=20) | Control Group (N=17)
Fracture left forearm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated
Acute gastroenteritis with dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated
Acute gastroenteritis with febrile seizure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated
Viral gastritis with dehydration/vomiting, fever (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Dengue Vaccine- 1/10 Dose (T-DEN F17 ) (N=4) | Cohort B: Full Dose (T-DEN F17 ) (N=10) | Cohort C: Dengue Vaccine - Full Dose (T-DEN F17 ) (N=20) | Control Group (N=17)
Pain (General disorders) | 1 (1) | 3 (3) | 8 (8) | 3 (3) — Dose 1
Redness (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (7) | 14 (14) | 1 (1) — Dose 1
Swelling (General disorders) | 1 (1) | 5 (5) | 11 (11) | 2 (2) — Dose 1
Pain (General disorders) | 1 (1) | 2 (2) | 11 (11) | 2 (2) — Dose 2
Redness (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 12 (12) | 3 (3) — Dose 2
Swelling (General disorders) | 1 (1) | 0 (0) | 8 (8) | 1 (1) — Dose 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No